CLINICAL TRIAL: NCT05399745
Title: BILACO Trial: Biliary Atresia - a Severe Complex Congenital Liver Disease With High Mortality, Compromised Neurological Development, Severe Malnutrition and Unknown Etiology
Brief Title: BILACO Trial: Biliary Atresia - a Severe Complex Congenital Liver Disease
Acronym: BILACO
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Brix Christensen, Principal investigator, MD, PhD, DMSc, senior consultant, Rigshospitalet, Denmark
Other Study IDs: H-19042934
Record Dates: First submitted 2022-03-08; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Biliary Atresia; Cognitive Impairment
MeSH Terms: conditions — Biliary Atresia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with biliary atresia
  Interventions: Other: Neurocognitive monitoring
- Children with Tetralogy of Fallot
  Interventions: Other: Neurocognitive monitoring
- Healthy control children
  Interventions: Other: Neurocognitive monitoring

INTERVENTIONS:
Other: Neurocognitive monitoring — Neurocognitive tests and MRI of the brain

SUMMARY:
Biliary atresia is the most severe form of cholestatic liver disease. The children have high morbidity and mortality and get devastating pruritus and fatigue, failure to thrive, progressive hepatic failure and impaired neurodevelopment. The etiology is mostly unknown. More than half need a new liver from a living or deceased donor during childhood. However, correct timing of the transplantation is extremely difficult because of lack of consensus based on clinical assessment tools. All though the incidence is low, the cost of this disease is tremendous from both a clinical and human perspective. So far, protocolized neurodevelopment tests, genetic profiling, precise malnutrition evaluation based on clinical appearance, biochemical markers and brain MRI-scans, body composition, immunological function, level of physical activity and optimal time of transplantation in cholestatic children are unknown.

The aim is to determine risk factors for neurocognitive impairment in children suffering from severe cholestasis in order to determine optimal time for liver transplantation from a brain perspective.

In a prospective study, the investigators will investigate risk factors related to brain-, heart-, gut- and immunological function in the Danish cohort. This cohort consists of 75 children aged 0-18 years. In addition, 30 aged and gender matched healthy and 20 tetra fallot children will serve as control groups. The children will undergo extensive and advanced liver function evaluation, genetic profiling, nutrition and immunological status, neuro-imaging and neurocognitive evaluation at time of diagnose, 2 years of age, pre-school, pre-teenage, and teenage. In case of a liver transplantation, additional neuro-cognitive tests will be performed

ELIGIBILITY:
Inclusion Criteria:

* Biliary atresia
* Tetralogy of Fallot
* Healthy controls

Exclusion Criteria:

- Not able to participate in exams

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with biliary atresia (BA), children with Tetralogy of Fallot (ToF) and healthy control children between the age of 0-17 years. The BA and ToF children were recruited from their respective outpatient clinics at Rigshospitalet, Denmark, which is the only centre treating these patients. Healthy controls were siblings to BA children, recruited from staffs children and friends or recruited from a general practitioners office in Nivaa, Denmark. The recruitment took place from March 2020 and is ongoing
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI of the brain | Inclusion
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive status: Early movement repertoire (General movement) | Inclusion
  Neurocognitive test panel depending on age at inclusion
  % of patients with of abnormal movement assessed using early movement repertoire (GM) if inclusion at diagnosis. Early movement repertoire is a measurement tool where abnormal movement is identified.
Neurocognitive status: Alberta Infant Motor Scale | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Alberta Infant Motor Scale if inclusion at diagnosis
  Percentile, highest is the best
Neurocognitive status: Bayley Scales of Development III | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Bayley Scales of Development III if inclusion up to 2.5 years:
  From 0-200, highest is best
Neurocognitive status: WIPPSI | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  WIPPSI if inclusion between 2.5-6 years:
  Wechsler Preschool and Primary Scale of Intelligence, from 41 to 160, highest is best
Neurocognitive status: ABC Movement | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  ABC Movement if inclusion between 2.5-16 years
  Movement Assessment Battery for Children, mean 10 SD 3, highest is best
Neurocognitive status: WISC-IV | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  WISC-IV if inclusion between 6-16 years
  Wechsler Intelligence Scale for Children, 40 to 160, highest is best
Neurocognitive status: Auditory Verbal Learning Test/ToMaL | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Auditory Verbal Learning Test/ToMaL if inclusion between 6-18 years Mean 10 SD 3, highest is best
Neurocognitive status: TEA-Ch | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  TEA-Ch if inclusion between 6-18 years
  Test of Everyday Attention for Children, normalized to z-score, highest is best
Neurocognitive status: BADS-C | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  BADS-C if inclusion between 6-18 years Behavioural Assessment of the Dysexecutive Syndrome in Children, 0-24, mean 10 SD 3, highest is best
Neurocognitive status: Test of Visual Perceptual Skills | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Test of Visual Perceptual Skills if inclusion between 6-18 years
  Percentile, highest is best
Neurocognitive status: CANTAB | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  CANTAB if inclusion between 6-18 years Cambridge Neuropsychological Test Automated Battery
Neurocognitive status: The Beery Visuo-Motor Integration test | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  The Beery Visuo-Motor Integration test if inclusion between 6-18 years Mean of 100 and standard deviation of 15, highest is best
Neurocognitive status: WAIS IV | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  WAIS IV if inclusion from 16 to 18 years Wechsler Adult Intelligence Scale, 40-160, highest is best
Neurocognitive status: Kiddie-sads | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Kiddie-sads if included between 2-18 years Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
Neurocognitive status: BRIEF 1 | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  BRIEF 1 if inclusion up to 6 years Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: BRIEF 2 | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  BRIEF 2 if inclusion between 6-18 years Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: CBCL | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  CBCL if included between 2-18 years Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: ADHD screening | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  ADHD screening if included between 2-18 years Lowest is best, 0-78
Neurocognitive status: SRS-2 | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  SRS-2 screening if included between 6-18 years
  Social Responsiveness Scale, 32-114. lowest is best
Neurocognitive status: Vineland | Inclusion
  Neurocognitive test panel depending on age at inclusion:
  Vineland screening if included between 6-18 years Vineland Adaptive Behavior Scales, 20 to 160, highest is best
MRI of the brain | 1 year
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive status: Alberta Infant Motor Scale | 1 year
  Alberta Infant Motor Scale Percentile, highest is the best
Neurocognitive status: Bayley Scales of Development III | 1 year
  Bayley Scales of Development III
  From 0-200, highest is best
Neurocognitive status: BRIEF 1 | 1 year
  BRIEF 1 Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: CBCL | 1 year
  CBCL Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: Kiddie-Sads | 1 year
  Kiddie-Sads Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
MRI of the brain | 2 years
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive status: Bayley Scales of Development III | 2 years
  Bayley Scales of Development III From 0-200, highest is best
Neurocognitive status: BRIEF 1 | 2 years
  BRIEF 1 Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: CBCL | 2 years
  CBCL Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: Kiddie-Sads | 2 years
  Kiddie-Sads Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
Neurocognitive status: ADHD | 2 years
  ADHD Lowest is best, 0-78
Neurocognitive status: Vineland | 2 years
  Vineland Adaptive Behavior Scales, 20 to 160, highest is best
MRI of the brain | 6 years
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive: Movement ABC | 6 years
  Neurocognitive test panel depending on age Movement Assessment Battery for Children, mean 10 SD 3, highest is best
Neurocognitive status: WISC-IV | 6 years
  WISC-IV
  Wechsler Intelligence Scale for Children, 40 to 160, highest is best
Neurocognitive status: Auditory Verbal Learning Test/ToMaL | 6 years
  Auditory Verbal Learning Test/ToMaL Mean 10 SD 3, highest is best
Neurocognitive status: TEA-Ch | 6 years
  TEA-Ch Test of Everyday Attention for Children, normalized to z-score, highest is best
Neurocognitive status: BADS-C | 6 years
  BADS-C Behavioural Assessment of the Dysexecutive Syndrome in Children, 0-24, mean 10 SD 3, highest is best
Neurocognitive status: Test of Visual Perceptual Skills | 6 years
  Test of Visual Perceptual Skills Percentile, highest is best
Neurocognitive status: The Beery Visuo-Motor Integration test | 6 years
  The Beery Visuo-Motor Integration test Mean of 100 and standard deviation of 15, highest is best
Neurocognitive status: CANTAB | 6 years
  CANTAB Cambridge Neuropsychological Test Automated Battery
Neurocognitive status: BRIEF 2 | 6 years
  BRIEF 2 Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: ADHD screening | 6 years
  ADHD screening Lowest is best, 0-78
Neurocognitive status: SRS-2 | 6 years
  SRS-2 Social Responsiveness Scale, 32-114. lowest is best
Neurocognitive status: Kiddie-Sads | 6 years
  Kiddie-Sads Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
Neurocognitive status: CBCL | 6 years
  CBCL Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: Vineland | 6 years
  Vineland Vineland Adaptive Behavior Scales, 20 to 160, highest is best
MRI of the brain | 11 years
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive status: Movement ABC | 11 years
  Neurocognitive test panel depending on age at inclusion:
  ABC Movement if inclusion between 2.5-16 years
  Movement Assessment Battery for Children, mean 10 SD 3, highest is best
Neurocognitive status: WISC-IV | 11 years
  WISC-IV
  Wechsler Intelligence Scale for Children, 40 to 160, highest is best
Neurocognitive status: Auditory Verbal Learning Test/ToMaL | 11 years
  Auditory Verbal Learning Test/ToMaL Mean 10 SD 3, highest is best
Neurocognitive status:TEA-Ch | 11 years
  TEA-Ch Test of Everyday Attention for Children, normalized to z-score, highest is best
Neurocognitive status: BADS-C | 11 years
  BADS-C Behavioural Assessment of the Dysexecutive Syndrome in Children, 0-24, mean 10 SD 3, highest is best
Neurocognitive status: Test of Visual Perceptual Skills | 11 years
  Test of Visual Perceptual Skills Percentile, highest is best
Neurocognitive status: The Beery Visuo-Motor Integration test | 11 years
  The Beery Visuo-Motor Integration test Mean of 100 and standard deviation of 15, highest is best
Neurocognitive status: CANTAB | 11 years
  CANTAB Cambridge Neuropsychological Test Automated Battery
Neurocognitive status: BRIEF 2 | 11 years
  BRIEF 2 Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: ADHD screening | 11 years
  ADHD screening Lowest is best, 0-78
Neurocognitive status: SRS-2 | 11 years
  SRS-2 Social Responsiveness Scale, 32-114. lowest is best
Neurocognitive status: Kiddie-Sads | 11 years
  Kiddie-Sads Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
Neurocognitive status: CBCL | 11 years
  CBCL Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: Vineland | 11 years
  Vineland Adaptive Behavior Scales, 20 to 160, highest is best
MRI of the brain | 16 years
  % of patients with anatomic anomalies on MRI of the brain
Neurocognitive status: Movement ABC | 16 years
  Neurocognitive test panel depending on age at inclusion:
  ABC Movement if inclusion between 2.5-16 years
  Movement Assessment Battery for Children, mean 10 SD 3, highest is best
Neurocognitive status: WISC-IV | 16 years
  WISC-IV Wechsler Adult Intelligence Scale, 40-160, highest is best
Neurocognitive status: Auditory Verbal Learning Test/ToMaL | 16 years
  Auditory Verbal Learning Test/ToMaL Mean 10 SD 3, highest is best
Neurocognitive status: TEA-Ch | 16 years
  TEA-Ch Test of Everyday Attention for Children, normalized to z-score, highest is best
Neurocognitive status: BADS-C | 16 years
  BADS-C Behavioural Assessment of the Dysexecutive Syndrome in Children, 0-24, mean 10 SD 3, highest is best
Neurocognitive status: Test of Visual Perceptual Skills | 16 years
  Test of Visual Perceptual Skills Percentile, highest is best
Neurocognitive status: The Beery Visuo-Motor Integration test | 16 years
  The Beery Visuo-Motor Integration test Mean of 100 and standard deviation of 15, highest is best
Neurocognitive status: CANTAB | 16 years
  CANTAB Cambridge Neuropsychological Test Automated Battery
Neurocognitive status: BRIEF 2 | 16 years
  BRIEF 2 Behaviour Rating Inventory of Executive Function, percentile, lowest is best
Neurocognitive status: ADHD screening | 16 years
  ADHD screening Lowest is best, 0-78
Neurocognitive status: SRS-2 | 16 years
  SRS-2 Social Responsiveness Scale, 32-114. lowest is best
Neurocognitive status: Kiddie-Sads | 16 years
  Kiddie-Sads Kiddie Schedule for Affective Disorders and Schizophrenia, 0-61, lowest is best
Neurocognitive status: CBCL | 16 years
  CBCL Child Behavior Checklist, percentile, lowest is best
Neurocognitive status: Vineland | 16 years
  Vineland Adaptive Behavior Scales, 20 to 160, highest is best

SECONDARY OUTCOMES:
Genetics: Whole genome sequencing of blood | Inclusion
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | Inclusion
  Whole genome sequencing of liver biopsy
Microbiome: Urine proteomics | Inclusion
  Microbiome measurements on urine
Microbiome: Feces proteomics | Inclusion
  Microbiome measurements on feces
Microbiome: Saliva proteomics | Inclusion
  Microbiome measurements on saliva
Microbiome: Feces Next Generation Sequencing of microbial DNA | Inclusion
  Microbiome measurement on feces
Microbiome: Urine Next Generation Sequencing of microbial DNA | Inclusion
  Microbiome measurement on urine
Microbiome: Saliva Next Generation Sequencing of microbial DNA | Inclusion
  Microbiome measurement on saliva
Microbiome: Feces metabolomics | Inclusion
  Microbiome measurements on feces
Microbiome: Urine metabolomics | Inclusion
  Microbiome measurements on urine
Microbiome: Saliva metabolomics | Inclusion
  Microbiome measurements on saliva
Microbiome: Feces metatranscriptomics | Inclusion
  Microbiome measurements on feces
Microbiome: Urine metatranscriptomics | Inclusion
  Microbiome measurements on urine
Microbiome: Saliva metatranscriptomics | Inclusion
  Microbiome measurements on saliva
Genetics: Whole genome sequencing of blood | 1 year
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | 1 year
  Whole genome sequencing of liver biopsy
Microbiome: Feces metatranscriptomics | 1 year
  Microbiome measurements on feces
Microbiome: Urine metatranscriptomics | 1 year
  Microbiome measurements on urine
Microbiome: Saliva metatranscriptomics | 1 year
  Microbiome measurements on saliva
Microbiome: Urine Next Generation Sequencing of microbial DNA | 1 year
  Microbiome measurements on urine
Microbiome: Feces Next Generation Sequencing of microbial DNA | 1 year
  Microbiome measurements on feces
Microbiome: Saliva Next Generation Sequencing of microbial DNA | 1 year
  Microbiome measurements on saliva
Microbiome: Saliva metabolomics | 1 year
  Microbiome measurements on saliva
Microbiome: Urine metabolomics | 1 year
  Microbiome measurements on urine
Microbiome: Feces metabolomics | 1 year
  Microbiome measurements on feces
Microbiome: Saliva proteomics | 1 year
  Microbiome measurements on saliva
Microbiome: Urine proteomics | 1 year
  Microbiome measurements on urine
Microbiome: Feces proteomics | 1 year
  Microbiome measurements on feces
Genetics: Whole genome sequencing of blood | 2 years
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | 2 years
  Whole genome sequencing of liver biopsy
Microbiome: Feces metatranscriptomics | 2 years
  Microbiome measurements on feces
Microbiome: Urine metatranscriptomics | 2 years
  Microbiome measurements on urine
Microbiome: Saliva metatranscriptomics | 2 years
  Microbiome measurements on saliva
Microbiome: Saliva metabolomics | 2 years
  Microbiome measurements on saliva
Microbiome: Feces metabolomics | 2 years
  Microbiome measurements on feces
Microbiome: Urine metabolomics | 2 years
  Microbiome measurements on urine
Microbiome: Urine proteomics | 2 years
  Microbiome measurements on urine
Microbiome: Feces proteomics | 2 years
  Microbiome measurements on feces
Microbiome: Saliva proteomics | 2 years
  Microbiome measurements on saliva
Microbiome: Urine Next Generation Sequencing of microbial DNA | 2 years
  Microbiome measurements on urine
Microbiome: Saliva Next Generation Sequencing of microbial DNA | 2 years
  Microbiome measurements on saliva
Microbiome: Feces Next Generation Sequencing of microbial DNA | 2 years
  Microbiome measurements on feces
Genetics: Whole genome sequencing of blood | 6 years
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | 6 years
  Whole genome sequencing of liver biopsy
Microbiome: Feces Next Generation Sequencing of microbial DNA | 6 years
  Microbiome measurements on feces
Microbiome: Feces metatranscriptomics | 6 years
  Microbiome measurements on feces
Microbiome: Feces metabolomics | 6 years
  Microbiome measurements on feces
Microbiome: Feces proteomics | 6 years
  Microbiome measurements on feces
Microbiome: Urine Next Generation Sequencing of microbial DNA | 6 years
  Microbiome measurements on urine
Microbiome: Urine metatranscriptomics | 6 years
  Microbiome measurements on urine
Microbiome: Urine metabolomics | 6 years
  Microbiome measurements on urine
Microbiome: Urine proteomics | 6 years
  Microbiome measurements on urine
Microbiome: Saliva Next Generation Sequencing of microbial DNA | 6 years
  Microbiome measurements on saliva
Microbiome: Saliva metatranscriptomics | 6 years
  Microbiome measurements on saliva
Microbiome: Saliva metabolomics | 6 years
  Microbiome measurements on saliva
Microbiome: Saliva proteomics | 6 years
  Microbiome measurements on saliva
Genetics: Whole genome sequencing of blood | 11 years
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | 11 years
  Whole genome sequencing of liver biopsy
Microbiome: Feces Next Generation Sequencing of microbial DNA | 11 years
  Microbiome measurements on feces
Microbiome: Feces metatranscriptomics | 11 years
  Microbiome measurements on feces
Microbiome: Feces metabolomics | 11 years
  Microbiome measurements on feces
Microbiome: Feces proteomics | 11 years
  Microbiome measurements on feces
Microbiome: Urine Next Generation Sequencing of microbial DNA | 11 years
  Microbiome measurements on urine
Microbiome: Urine metatranscriptomics | 11 years
  Microbiome measurements on urine
Microbiome: Urine metabolomics | 11 years
  Microbiome measurements on urine
Microbiome: Urine proteomics | 11 years
  Microbiome measurements on urine
Microbiome: Saliva Next Generation Sequencing of microbial DNA | 11 years
  Microbiome measurements on saliva
Microbiome: Saliva metatranscriptomics | 11 years
  Microbiome measurements on saliva
Microbiome: Saliva metabolomics | 11 years
  Microbiome measurements on saliva
Microbiome: Saliva proteomics | 11 years
  Microbiome measurements on saliva
Genetics: Whole genome sequencing of blood | 16 years
  Whole genome sequencing of blood
Genetics: Whole genome sequencing of liver biopsy | 16 years
  Whole genome sequencing of liver biopsy
Microbiome: Feces metatranscriptomics | 16 years
  Microbiome measurements on feces
Microbiome: Feces Next Generation Sequencing of microbial DNA | 16 years
  Microbiome measurements on feces
Microbiome: Feces metabolomics | 16 years
  Microbiome measurements on feces
Microbiome: Feces proteomics | 16 years
  Microbiome measurements on feces
Microbiome: Urine metatranscriptomics | 16 years
  Microbiome measurements on urine
Microbiome: Urine Next Generation Sequencing of microbial DNA | 16 years
  Microbiome measurements on urine
Microbiome: Urine metabolomics | 16 years
  Microbiome measurements on urine
Microbiome: Urine proteomics | 16 years
  Microbiome measurements on urine
Microbiome: Saliva metatranscriptomics | 16 years
  Microbiome measurements on saliva
Microbiome: Saliva Next Generation Sequencing of microbial DNA | 16 years
  Microbiome measurements on saliva
Microbiome: Saliva metabolomics | 16 years
  Microbiome measurements on saliva
Microbiome: Saliva proteomics | 16 years
  Microbiome measurements on saliva
Status of the cardiac system: Ultrasound of the heart | Inclusion
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | Inclusion
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | Inclusion
  Near Infrared Fluorescence of the lymph system
Status of the cardiac system: Ultrasound of the heart | 1 year
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | 1 year
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | 1 year
  Near Infrared Fluorescence of the lymph system
Status of the cardiac system: Ultrasound of the heart | 2 years
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | 2 years
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | 2 years
  Near Infrared Fluorescence of the lymph system
Status of the cardiac system: Ultrasound of the heart | 6 years
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | 6 years
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | 6 years
  Near Infrared Fluorescence of the lymph system
Status of the cardiac system: Ultrasound of the heart | 11 years
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | 11 years
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | 11 years
  Near Infrared Fluorescence of the lymph system
Status of the cardiac system: Ultrasound of the heart | 16 years
  % of patients with anatomic anomalies on ultrasound of the heart
Status of the cardiac system: MRI of the lymph system | 16 years
  % of patients with central lymph system anomaly
Status of the cardiac system: Near Infrared Fluorescence of the lymph system | 16 years
  Near Infrared Fluorescence of the lymph system
Level of Physical activity | Inclusion
  Accelerometer measurements
Level of Physical activity | 1 year
  Accelerometer measurements
Level of Physical activity | 2 years
  Accelerometer measurements
Level of Physical activity | 6 years
  Accelerometer measurements
Level of Physical activity | 11 years
  Accelerometer measurements
Level of Physical activity | 16 years
  Accelerometer measurements
Ultrasound of liver and bile ducts with elastography | Inclusion
  % of patients with liver fibrosis measured with ultrasound
Liver biopsy | Inclusion
  Level of liver fibrosis (grade 0-4)
FGF-19; Fibroblast growth factor 19 | Inclusion
  Liver fibrosis status
ELF-score: Enhanced Liver Fibrosis | Inclusion
  Liver fibrosis status
INR: international normalized ratio | Inclusion
  Standard liver evaluation
prothrombin+proconvertin (PP) | Inclusion
  Standard liver evaluation
ALAT: alanine transaminase | Inclusion
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | Inclusion
  Standard liver evaluation
Bilirubin | Inclusion
  Standard liver evaluation
ASAT: Aspartate transaminase | Inclusion
  Standard liver evaluation
Alkaline phosphatase | Inclusion
  Standard liver evaluation
Ammonia | Inclusion
  Standard liver evaluation
Thrombocytes | Inclusion
  Standard liver evaluation
Ultrasound of liver and bile ducts with elastography | 1 year
  % of patients with liver fibrosis measured with ultrasound
FGF-19: Fibroblast growth factor 19 | 1 year
  Liver fibrosis status
ELF-score: Enhanced Liver Fibrosis | 1 year
  Liver fibrosis status
INR: international normalized ratio | 1 year
  Standard liver evaluation
prothrombin+proconvertin (PP) | 1 year
  Standard liver evaluation
ALAT: alanine transaminase | 1 year
  Standard liver evaluation
ASAT: Aspartate transaminase | 1 year
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | 1 year
  Standard liver evaluation
Bilirubin | 1 year
  Standard liver evaluation
Alkaline phosphatase | 1 year
  Standard liver evaluation
Ammonia | 1 year
  Standard liver evaluation
Thrombocytes | 1 year
  Standard liver evaluation
Liver biopsy | 1 year
  Level of liver fibrosis (grade 0-4)
Ultrasound of liver and bile ducts with elastography | 2 years
  % of patients with liver fibrosis measured with ultrasound
FGF-19: Fibroblast growth factor 19 | 2 years
  Liver fibrosis status
ELF-score: Enhanced Liver Fibrosis | 2 years
  Liver fibrosis status
Liver biopsy | 2 years
  Level of liver fibrosis (grade 0-4)
INR: international normalized ratio | 2 years
  Standard liver evaluation
prothrombin+proconvertin (PP) | 2 years
  Standard liver evaluation
ALAT: alanine transaminase | 2 years
  Standard liver evaluation
ASAT: Aspartate transaminase | 2 years
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | 2 years
  Standard liver evaluation
Alkaline phosphatase | 2 years
  Standard liver evaluation
Bilirubin | 2 years
  Standard liver evaluation
Ammonia | 2 years
  Standard liver evaluation
Thrombocytes | 2 years
  Standard liver evaluation
Ultrasound of liver and bile ducts with elastography | 6 years
  % of patients with liver fibrosis measured with ultrasound
Liver biopsy | 6 years
  Level of liver fibrosis (grade 0-4)
ELF-score: Enhanced Liver Fibrosis | 6 years
  Liver fibrosis status
FGF-19: Fibroblast growth factor 19 | 6 years
  Liver fibrosis status
INR: international normalized ratio | 6 years
  Standard liver evaluation
prothrombin+proconvertin (PP) | 6 years
  Standard liver evaluation
ALAT: alanine transaminase | 6 years
  Standard liver evaluation
ASAT: Aspartate transaminase | 6 years
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | 6 years
  Standard liver evaluation
Bilirubin | 6 years
  Standard liver evaluation
Alkaline phosphatase | 6 years
  Standard liver evaluation
Ammonia | 6 years
  Standard liver evaluation
Thrombocytes | 6 years
  Standard liver evaluation
Ultrasound of liver and bile ducts with elastography | 11 years
  % of patients with liver fibrosis measured with ultrasound
Liver biopsy | 11 years
  Level of liver fibrosis (grade 0-4)
FGF-19: Fibroblast growth factor 19 | 11 years
  Liver fibrosis status
ELF-score: Enhanced Liver Fibrosis | 11 years
  Liver fibrosis status
INR: international normalized ratio | 11 years
  Standard liver evaluation
prothrombin+proconvertin (PP) | 11 years
  Standard liver evaluation
ALAT: alanine transaminase | 11 years
  Standard liver evaluation
ASAT: Aspartate transaminase | 11 years
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | 11 years
  Standard liver evaluation
Bilirubin | 11 years
  Standard liver evaluation
Alkaline phosphatase | 11 years
  Standard liver evaluation
Ammonia | 11 years
  Standard liver evaluation
Thrombocytes | 11 years
  Standard liver evaluation
Ultrasound of liver and bile ducts with elastography | 16 years
  % of patients with liver fibrosis measured with ultrasound
Liver biopsy | 16 years
  Level of liver fibrosis (grade 0-4)
FGF-19: Fibroblast growth factor 19 | 16 years
  Liver fibrosis status
ELF-score: Enhanced Liver Fibrosis | 16 years
  Liver fibrosis status
INR: international normalized ratio | 16 years
  Standard liver evaluation
prothrombin+proconvertin (PP) | 16 years
  Standard liver evaluation
ALAT: alanine transaminase | 16 years
  Standard liver evaluation
ASAT: Aspartate transaminase | 16 years
  Standard liver evaluation
GGT: Gamma-glutamyl transferase | 16 years
  Standard liver evaluation
Bilirubin | 16 years
  Standard liver evaluation
Alkaline phosphatase | 16 years
  Standard liver evaluation
Ammonia | 16 years
  Standard liver evaluation
Thrombocytes | 16 years
  Standard liver evaluation
Clinical examination: Cirrhosis stigmata | Inclusion
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | 1 year
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | 2 years
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | 6 years
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | 11 years
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | 16 years
  Incidence of spider angioma
Clinical examination: Cirrhosis stigmata | Inclusion
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | 1 year
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | 2 years
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | 6 years
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | 11 years
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | 16 years
  Incidence of ascitis
Clinical examination: Cirrhosis stigmata | Inclusion
  Incidence of palmar erythema
Clinical examination: Cirrhosis stigmata | 1 year
  Incidence of palmar erythema
Clinical examination: Cirrhosis stigmata | 2 years
  Incidence of palmar erythema
Clinical examination: Cirrhosis stigmata | 6 years
  Incidence of palmar erythema
Clinical examination: Cirrhosis stigmata | 11 years
  Incidence of palmar erythema
Clinical examination: Cirrhosis stigmata | 16 years
  Incidence of palmar erythema
Anthropometry: Length | Inclusion
  cm
Anthropometry: Length | 1 year
  cm
Anthropometry: Length | 2 years
  cm
Anthropometry: Height | 6 years
  cm
Anthropometry: Height | 11 years
  cm
Anthropometry: Height | 16 years
  cm
Anthropometry: Weight | Inclusion
  kg
Anthropometry: Weight | 1 year
  kg
Anthropometry: Weight | 2 years
  kg
Anthropometry: Weight | 6 years
  kg
Anthropometry: Weight | 11 years
  kg
Anthropometry: Weight | 16 years
  kg
Anthropometry: Mid-upper arm circumference (MUAC) | Inclusion
  mm
Anthropometry: Mid-upper arm circumference (MUAC) | 1 year
  mm
Anthropometry: Mid-upper arm circumference (MUAC) | 2 years
  mm
Anthropometry: Mid-upper arm circumference (MUAC) | 6 years
  mm
Anthropometry: Mid-upper arm circumference (MUAC) | 11 years
  mm
Anthropometry: Mid-upper arm circumference (MUAC) | 16 years
  mm
Anthropometry: Head circumference | Inclusion
  cm
Anthropometry: Head circumference | 1 year
  cm
Anthropometry: Head circumference | 2 years
  cm
Anthropometry: Head circumference | 6 years
  cm
Anthropometry: Head circumference | 11 years
  cm
Anthropometry: Head circumference | 16 years
  cm
Essential fatty acids | Inclusion
Essential fatty acids | 1 year
Essential fatty acids | 2 years
Essential fatty acids | 6 years
Essential fatty acids | 11 years
Essential fatty acids | 16 years
IGF-1 | Inclusion
  Insulin-like growth factor 1
IGF-1 | 1 year
  Insulin-like growth factor 1
IGF-1 | 2 years
  Insulin-like growth factor 1
IGF-1 | 6 years
  Insulin-like growth factor 1
IGF-1 | 11 years
  Insulin-like growth factor 1
IGF-1 | 16 years
  Insulin-like growth factor 1
Meal stimulation measuring incretin | Inclusion
Meal stimulation measuring incretin | 1 year
Meal stimulation measuring incretin | 2 years
Meal stimulation measuring incretin | 6 years
Meal stimulation measuring incretin | 11 years
Meal stimulation measuring incretin | 16 years
Bile acid | Inclusion
Bile acid | 1 year
Bile acid | 2 years
Bile acid | 6 years
Bile acid | 11 years
Bile acid | 16 years
Autotaxin | Inclusion
Autotaxin | 1 year
Autotaxin | 2 years
Autotaxin | 6 years
Autotaxin | 11 years
Autotaxin | 16 years
EDTA clearance | Inclusion
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
EDTA clearance | 1 year
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
EDTA clearance | 2 years
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
EDTA clearance | 6 years
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
EDTA clearance | 11 years
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
EDTA clearance | 16 years
  Glomerular Filtration Rate Measured by 51 Cr-EDTA Clearance
Vaccination status | Inclusion
  Level of antibodies
Vaccination status | 1 year
  Level of antibodies
Vaccination status | 2 years
  Level of antibodies
Vaccination status | 6 years
  Level of antibodies
Vaccination status | 11 years
  Level of antibodies
Vaccination status | 16 years
  Level of antibodies
Immunoresponse: RTE | Inclusion
  Recent thymic emigrants
Immunoresponse: RTE | 1 year
  Recent thymic emigrants
Immunoresponse: RTE | 2 years
  Recent thymic emigrants
Immunoresponse: RTE | 6 years
  Recent thymic emigrants
Immunoresponse: RTE | 11 years
  Recent thymic emigrants
Immunoresponse: RTE | 16 years
  Recent thymic emigrants
Immunoresponse: Flow panel | Inclusion
  T-cell differentiation
Immunoresponse: Flow panel | 1 year
  T-cell differentiation
Immunoresponse: Flow panel | 2 years
  T-cell differentiation
Immunoresponse: Flow panel | 6 years
  T-cell differentiation
Immunoresponse: Flow panel | 11 years
  T-cell differentiation
Immunoresponse: Flow panel | 16 years
  T-cell differentiation
Immunoresponse: Immunoglobulin | Inclusion
Immunoresponse: Immunoglobulin | 1 year
Immunoresponse: Immunoglobulin | 2 years
Immunoresponse: Immunoglobulin | 6 years
Immunoresponse: Immunoglobulin | 11 years
Immunoresponse: Immunoglobulin | 16 years
Immunoresponse: Somatic hyper mutation | Inclusion
Immunoresponse: Somatic hyper mutation | 1 year
Immunoresponse: Somatic hyper mutation | 2 years
Immunoresponse: Somatic hyper mutation | 6 years
Immunoresponse: Somatic hyper mutation | 11 years
Immunoresponse: Somatic hyper mutation | 16 years
Epstein-Barr Virus (EBV) | Inclusion
  level of EBV DNA present
Epstein-Barr Virus (EBV) | 1 year
  level of EBV DNA present
Epstein-Barr Virus (EBV) | 2 years
  level of EBV DNA present
Epstein-Barr Virus (EBV) | 6 years
  level of EBV DNA present
Epstein-Barr Virus (EBV) | 11 years
  level of EBV DNA present
Epstein-Barr Virus (EBV) | 16 years
  level of EBV DNA present
Cytomegalovirus (CMV) | Inclusion
  level of CMV DNA present
Cytomegalovirus (CMV) | 1 year
  level of CMV DNA present
Cytomegalovirus (CMV) | 2 years
  level of CMV DNA present
Cytomegalovirus (CMV) | 6 years
  level of CMV DNA present
Cytomegalovirus (CMV) | 11 years
  level of CMV DNA present
Cytomegalovirus (CMV) | 16 years
  level of CMV DNA present
Hepatobiliary scintigraphy | Inclusion
  Hepatic extraction fraction
Hepatobiliary scintigraphy | 1 year
  Hepatic extraction fraction
Hepatobiliary scintigraphy | 2 years
  Hepatic extraction fraction
Hepatobiliary scintigraphy | 6 years
  Hepatic extraction fraction
Hepatobiliary scintigraphy | 11 years
  Hepatic extraction fraction
Hepatobiliary scintigraphy | 16 years
  Hepatic extraction fraction
MRI of liver and bile ducts with elastography | Inclusion
  Liver stiffness
MRI of liver and bile ducts with elastography | 1 year
  Liver stiffness
MRI of liver and bile ducts with elastography | 2 years
  Liver stiffness
MRI of liver and bile ducts with elastography | 6 years
  Liver stiffness
MRI of liver and bile ducts with elastography | 11 years
  Liver stiffness
MRI of liver and bile ducts with elastography | 16 years
  Liver stiffness
Fibroscan | Inclusion
  Liver stiffness (number)
Fibroscan | 1 year
  Liver stiffness (number)
Fibroscan | 2 years
  Liver stiffness (number)
Fibroscan | 6 years
  Liver stiffness (number)
Fibroscan | 11 years
  Liver stiffness (number)
Fibroscan | 16 years
  Liver stiffness (number)
Indocyanine green clearance | Inclusion
Indocyanine green clearance | 1 year
Indocyanine green clearance | 2 years
Indocyanine green clearance | 6 years
Indocyanine green clearance | 11 years
Indocyanine green clearance | 16 years
Fecal fat measurements | Inclusion
Fecal fat measurements | 1 year
Fecal fat measurements | 2 years
Fecal fat measurements | 6 years
Fecal fat measurements | 11 years
Fecal fat measurements | 16 years
Thymus scan with ultrasound | Inclusion
  Thymic index (measurement of size)
Thymus scan with ultrasound | 1 year
  Thymic index (measurement of size)
Thymus scan with ultrasound | 2 years
  Thymic index (measurement of size)
Thymus scan with ultrasound | 6 years
  Thymic index (measurement of size)
Thymus scan with ultrasound | 11 years
  Thymic index (measurement of size)
Thymus scan with ultrasound | 16 years
  Thymic index (measurement of size)
DEXA scan | Inclusion
  Dual energy x-ray absorptiometry
DEXA scan | 1 year
  Dual energy x-ray absorptiometry
DEXA scan | 2 years
  Dual energy x-ray absorptiometry
DEXA scan | 6 years
  Dual energy x-ray absorptiometry
DEXA scan | 11 years
  Dual energy x-ray absorptiometry
DEXA scan | 16 years
  Dual energy x-ray absorptiometry
PEDS-QL | Inclusion
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
PEDS-QL | 1 year
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
PEDS-QL | 2 years
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
PEDS-QL | 6 years
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
PEDS-QL | 11 years
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
PEDS-QL | 16 years
  Pediatric Quality of Life Inventory Higher scores indicate better quality of life, from 0-100
Leptin | Inclusion
Leptin | 1 year
Leptin | 2 years
Leptin | 6 years
Leptin | 11 years
Leptin | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Brix Christensen, MD, PhD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No allowed from Danish government